CLINICAL TRIAL: NCT02508870
Title: A Phase Ib Study of the Safety and Pharmacology of Atezolizumab (Anti-PD-L1 Antibody) Administered Alone or in Combination With Azacitidine in Patients With Myelodysplastic Syndromes
Brief Title: A Study of Atezolizumab Administered Alone or in Combination With Azacitidine in Participants With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29754
Record Dates: First submitted 2015-07-24; First posted 2015-07-27 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — atezolizumab; Azacitidine

ARMS (6):
- Cohort A: Atezolizumab - HMA R/R MDS (Experimental): Participants with MDS who are HMA R/R will receive atezolizumab 1200 milligrams (mg) intravenous (IV) infusion every 3 weeks (Q3W) (21-day cycle). Treatment will continue for up to 17 cycles or until loss of clinical benefit, evidence of unacceptable toxicity, non-compliance with the protocol, voluntary withdrawal from the study, or study termination, whichever occurs first. Participants who achieve/maintain a partial response (PR) or hematological improvement (HI) after receiving 17 cycles of therapy may continue on study treatment beyond Cycle 17 until loss of clinical benefit.
  Interventions: Drug: Atezolizumab
- Cohort B: Atezolizumab+Azacitidine - HMA R/R MDS (Experimental): Induction: Participants with MDS who are HMA R/R will receive atezolizumab 840 mg IV infusion on Days 8 and 22 of each 28-day cycle along with azacitidine 75 milligrams per square meter (mg/m^2) subcutaneously (SC) on Days 1 to 7 of 28-day cycle, for 6 cycles. Maintenance: Participants who complete induction treatment will receive atezolizumab 1200 mg IV infusion Q3W (21-day cycle) for up to 8 additional cycles. Participants who achieve/maintain a PR or HI after completing the 8 cycles of atezolizumab maintenance therapy, may continue on study treatment until loss of clinical benefit.
  Interventions: Drug: Atezolizumab; Drug: Azacitidine
- Cohort C1: Atezolizumab+Azacitidine - HMA-Naive MDS (Experimental): Participants with MDS who are HMA-naive will receive atezolizumab 840 mg IV infusion on Days 8 and 22 of each 28-day cycle along with azacitidine 75 mg/m^2 SC on Days 1 to 7 of 28-day cycle, until loss of clinical benefit, evidence of unacceptable toxicity, non-compliance with the protocol, voluntary withdrawal from the study, or study termination, whichever occurs first.
  Interventions: Drug: Atezolizumab; Drug: Azacitidine
- Cohort C2: Atezolizumab+Azacitidine - HMA-Naive MDS (Experimental): If the participants enrolled in Cohort C1 fulfil the dose limiting toxicity (DLT) criteria, then additional participants with MDS who are HMA-naïve will receive atezolizumab 840 mg IV infusion on Days 8 and 22 of each 28-day cycle along with azacitidine 75 mg/m^2 SC on Days 1 to 7 of 28-day cycle, until loss of clinical benefit, evidence of unacceptable toxicity, non-compliance with the protocol, voluntary withdrawal from the study, or study termination, whichever occurs first.
  Interventions: Drug: Atezolizumab; Drug: Azacitidine
- Cohort A2: Atezolizumab - HMA R/R MDS (Experimental): If atezolizumab alone or in combination with azacitidine is found to be initially safe and tolerable in participants with HMA R/R MDS in both Cohorts A and B, then additional randomly assigned participants will receive atezolizumab 1200 mg IV infusion Q3W (21-day cycle). Treatment will continue for up to 17 cycles or until loss of clinical benefit, evidence of unacceptable toxicity, non-compliance with the protocol, voluntary withdrawal from the study, or study termination, whichever occurs first. Participants who achieve/maintain a PR or HI after receiving 17 cycles of therapy may continue on study treatment beyond Cycle 17 until loss of clinical benefit.
  Interventions: Drug: Atezolizumab
- Cohort B2: Atezolizumab+Azacitidine - HMA R/R MDS (Experimental): If atezolizumab alone or in combination with azacitidine is found to be initially safe and tolerable in participants with HMA R/R MDS in both Cohorts A and B, then additional randomly assigned participants will receive atezolizumab 840 mg IV infusion on Days 8 and 22 of each 28-day cycle along with azacitidine 75 mg/m^2 SC on Days 1 to 7 of 28-day cycle, for 6 cycles during induction. Participants who complete induction treatment will receive maintenance atezolizumab 1200 mg IV infusion Q3W (21-day cycle) for up to 8 additional cycles. Participants who achieve/maintain a PR or HI after completing the 8 cycles of atezolizumab maintenance therapy, may continue on study treatment until loss of clinical benefit.
  Interventions: Drug: Atezolizumab; Drug: Azacitidine

INTERVENTIONS:
Drug: Atezolizumab — Participants will receive atezolizumab as per the schedule described in individual cohort.
  Other Names: Tecentriq; MPDL3280A; RO5541267
Drug: Azacitidine — Participants will receive azacitidine as per the schedule described in individual cohort.
  Other Names: Vidaza
  Arms: Cohort B2: Atezolizumab+Azacitidine - HMA R/R MDS; Cohort B: Atezolizumab+Azacitidine - HMA R/R MDS; Cohort C1: Atezolizumab+Azacitidine - HMA-Naive MDS; Cohort C2: Atezolizumab+Azacitidine - HMA-Naive MDS

SUMMARY:
This is a multicenter, open-label, Phase 1b study of atezolizumab (anti-programmed death-ligand 1 [anti-PD-L1] monoclonal antibody) in participants who have hypomethylating agent (HMA)-naïve myelodysplastic syndromes (MDS) and are International Prognostic Scoring System-Revised (IPSS-R) intermediate/high/very high-risk, or have MDS relapsed or are refractory (R/R) to prior HMA therapy. The primary objectives of this study are to determine the safety and tolerability of atezolizumab therapy in these participant populations, including treatment in combination with azacitidine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDS (participants with therapy-related MDS are eligible)
* Eastern Cooperative Oncology Group (ECOG) performance status score less than or equal to (</=) 2
* Adequate end-organ function, as determined by laboratory tests obtained within 28 days prior to the first dose of study drug
* Willing and able to undergo a pre-treatment bone marrow biopsy and subsequent on-treatment bone marrow biopsies
* Women who are not postmenopausal or surgically sterile must have a negative serum pregnancy test result within 28 days prior to initiation of study drug
* For women of childbearing potential and men: agreement to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive measures

For participants in Cohorts A, A2, B, and B2:

* Progression at any time after initiation of azacitidine or decitabine treatment OR
* Failure to achieve complete or partial response or hematological improvement after at least six 4-week cycles of azacitidine or either four 4-week or four 6-week cycles of decitabine OR
* Relapse after initial complete or partial response or hematological improvement after six 4-week cycles of azacitidine or either four 4-week or four 6-week cycles of decitabine administered within the past 2 years

For participants in Cohorts C1 and C2:

* Must not have received prior treatment for MDS with any hypomethylating agent
* IPSS-R risk category of Intermediate, High, or Very High assessed at screening

Exclusion Criteria:

* Participants with a diagnosis of MDS secondary to paroxysmal nocturnal hemoglobinuria (PNH), aplastic anemia, or another inherited bone marrow failure disorder
* Prior allogeneic stem cell transplant or solid organ transplant
* Pregnant or lactating, or intending to become pregnant during the study
* Investigational therapy within 28 days prior to initiation of study treatment
* Immunosuppressive therapy within 6 weeks of Cycle 1, Day 1
* Prior treatment with immune checkpoint blockade therapies (anti-cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], anti-programmed death-1 [PD-1] or anti-PD-L1) or immune agonists (anti-cluster of differentiation [CD] 137, anti-CD40, anti-OX40)
* Any other therapy or serious medical condition, as specified in the protocol, or abnormality in clinical laboratory tests that, in the investigator's judgement, precludes the participant's safe participation in and completion of the study
* Left ventricular ejection fraction (LVEF) </= 40 percent (%) at screening
* Planned major surgery during the study or within 4 weeks of Cycle 1, Day 1
* History of idiopathic pulmonary fibrosis, organizing pneumonitis, drug-induced pneumonitis, or idiopathic pneumonitis or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with DLTs | Cohort A: Days 1 to 21; Cohorts B and C1: Days 1 to 28
Recommended Phase 2 Dose (RP2D) of Atezolizumab in Combination with Azacitidine | Cohort A: Days 1 to 21; Cohorts B and C1: Days 1 to 28
Percentage of Participants with Adverse Events (AEs) | Baseline up to approximately 3.5 years

SECONDARY OUTCOMES:
Cohorts A and A2: Percentage of Participants with Anti-Drug Antibodies (ADAs) to Atezolizumab | Pre-infusion (0 hour [0h]) on Day 1 (D1) of Cycles (Cy) 1, 2, 3, 4, 8, 12, and 16, end of treatment (EOT) (up to approximately 3.5 years [Yr]), and 90 days after last dose (up to approximately 3.5 Yr) (Cy length = 21 days)
Cohorts B and B2: Percentage of Participants with ADAs to Atezolizumab | Pre-infusion (0h) on Cy1, 2 Days 8 (D8) & 22 (D22) & Cy3 D8; pre-infusion (0h) on Cy7 D1 & then every 8 Cy up to EOT (approximately 3.5 Yr) and 90 days after last dose (approximately 3.5 Yr) (Cy length = 21 or 28 days)
Cohorts C1 and C2: Percentage of Participants with ADAs to Atezolizumab | Pre-infusion (0h) on Cy1, 2 D8 & D22 & Cy3 D8; pre-infusion (0h) on Cy7 D8 & then every 8 Cy up to EOT (approximately 3.5 Yr) and 90 days after last dose (approximately 3.5 Yr) (Cy length = 21 or 28 days)
Cohorts A and A2: Maximum Serum Concentration (Cmax) of Atezolizumab | Pre-infusion (0h), 30 minutes (min) post 60-min infusion on Cy 1 D1; pre-infusion (0h) on D1 of Cy 2, 3, 4, 8, 12, & 16, EOT (approximately 3.5 Yr); 90 days after EOT (approximately 3.5 Yr) (Cy length = 21 days)
Cohorts B and B2: Cmax of Atezolizumab | Pre-infusion (0h), 30 min post 60-min infusion on Cy1D8; pre-infusion (0h) on Cy1D22, Cy2D8 & 22, Cy3D8, Cy7D1, every 8 Cy up to EOT (approximately 3.5 Yr); 90 days after EOT (approximately 3.5 Yr) (1 Cy = 21 or 28 days)
Cohorts C1 and C2: Cmax of Atezolizumab | Pre-infusion (0h), 30 min post 60-min infusion on Cy1D8; pre-infusion (0h) on Cy1D22, Cy2D8 & 22, Cy3D8, Cy7D8, every 8 Cy up to EOT (approximately 3.5 Yr); 90 days after EOT (approximately 3.5 Yr) (1 Cy = 21 or 28 days)
Cohorts A and A2: Minimum Serum Concentration (Cmin) of Atezolizumab | Pre-infusion (0h), 30 minutes (min) post 60-min infusion on Cy 1 D1; pre-infusion (0h) on D1 of Cy 2, 3, 4, 8, 12, & 16, EOT (approximately 3.5 Yr); 90 days after EOT (approximately 3.5 Yr) (Cy length = 21 days)
Cohorts B and B2: Cmin of Atezolizumab | Pre-infusion (0h), 30 min post 60-min infusion on Cy1D8; pre-infusion (0h) on Cy1D22, Cy2D8 & 22, Cy3D8, Cy7D1, every 8 Cy up to EOT (approximately 3.5 Yr); 90 days after EOT (approximately 3.5 Yr) (1 Cy = 21 or 28 days)
Cohorts C1 and C2: Cmin of Atezolizumab | Pre-infusion (0h), 30 min post 60-min infusion on Cy1D8; pre-infusion (0h) on Cy1D22, Cy2D8 & 22, Cy3D8, Cy7D8, every 8 Cy up to EOT (approximately 3.5 Yr); 90 days after EOT (approximately 3.5 Yr) (1 Cy = 21 or 28 days)
Percentage of Participants with Overall Response, According to 2006 International Working Group (IWG) Response Criteria for MDS | Randomization up to disease progression or death, whichever occurs first (up to approximately 3.5 years)
Percentage of Participants with Overall Response After Induction Therapy, According to 2006 IWG Response Criteria for MDS | After end of induction up to disease progression or death, whichever occurs first (up to approximately 3.5 years)
Duration of Clinical Response, According to 2006 IWG Response Criteria for MDS | Time from the initial overall response to the time of disease progression or death, whichever occurs first (up to approximately 3.5 years)
Time to Acute Myeloid Leukemia (AML) Progression, According to 2006 IWG Response Criteria for MDS | Randomization up to the date of AML progression (up to approximately 3.5 years)
Progression Free Survival (PFS), According to 2006 IWG Response Criteria for MDS | Randomization up to disease progression or death, whichever occurs first (up to approximately 3.5 years)
Cohorts A, A2, B, and B2: Overall Survival (OS) | Randomization up to death due to any cause (up to approximately 3.5 years)
Percentage of Participants With Change in Red Cell and Platelet Transfusion | Baseline up to approximately 3.5 years
Cohorts A2 or B2: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Score | D1 of every Cy up to study discontinuation (approximately 3.5 Yr) (1 Cy = 21 or 28 days)
Cohorts A2 and B2: Functional Assessment of Chronic Illness Therapy Fatigue Questionnaire (FACIT-Fatigue) Score | D1 of every Cy up to study discontinuation (approximately 3.5 Yr) (1 Cy = 21 or 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- United States (15):
  - City of Hope, Duarte, California
  - Stanford University, Palo Alto, California
  - University of California, San Francisco, Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Kansas Medical Center, Westwood, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Nebraska Medical Center; UNMC Oncology/Hematology, Omaha, Nebraska
  - Roswell Park Cancer Institute; Grace Cancer Drug Center, Buffalo, New York
  - Montefiore Einstein Cancer Center, The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Medical University of South Carolina; Hollings Cancer Center, Charleston, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Health System; Hematology/Oncology Division, Charlottesville, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Gerds AT, Scott BL, Greenberg P, Lin TL, Pollyea DA, Verma A, Dail M, Feng Y, Green C, Ma C, Medeiros BC, Yan M, Yousefi K, Donnellan W. Atezolizumab alone or in combination did not demonstrate a favorable risk-benefit profile in myelodysplastic syndrome. Blood Adv. 2022 Feb 22;6(4):1152-1161. doi: 10.1182/bloodadvances.2021005240. PMID 34932793